CLINICAL TRIAL: NCT05504824
Title: The Effect of Case-Based Education on the Development of Nursing Students' Clinical Reasoning Skills in Critical Illness: A Pilot Randomized Controlled Trial
Brief Title: The Effect of Case-Based Education on the Development of Nursing Students' Clinical Reasoning Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ayşegül Öztürk Birge, Assistant Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AU-OBIRGE-001
Record Dates: First submitted 2022-08-04; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Clinical Reasoning; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Students in both experimental groups were applied the student information form and the pretest of the CRCF between May 18 and 20, 2021 before the education. The schedule of the education intervention was determined according to the convenience of the students in the experimental group. Accordingly, the experimental group was given education between June 8 and 11, 2021. After the education sessions were completed, experimental groups were applied the CRCF as a posttest on June 28, 2021. The students in the experimental group were asked to fill out the "Student Satisfaction with Education Questionnaire" and the "Form for Views on the Education" online.
  Interventions: Other: Case-based education
- Control group (No Intervention): Students in control groups were applied the student information form and the pretest of the CRCF between May 18 and 20, 2021 before the education. The students in the control group continued their current standard education process. After the education sessions were completed, control groups were applied the CRCF as a posttest on June 28, 2021.

INTERVENTIONS:
Other: Case-based education — The education phase This stage included the explanation of the CR process, the analysis of CR cases, the drafting of new cases suitable for the CR process by students, and the analysis process.
  The education program was carried out on a web platform (Zoom) consistent with the changes in the COVID-19 pandemic process. The CR cases to be used in case-based education were sent to the students via e-mail before the group interview to make sure students came prepared for the group discussion. In case-based education, after the students read the case, they were asked some questions to determine their decisions and reasoning.
  Arms: Experimental group

SUMMARY:
Aim: This study was conducted to determine the effect of case-based education on the development of clinical reasoning skills of nursing students in critical illnesses.

Methods: The study was conducted between January 20 and June 30, 2021 using a pilot randomized controlled trial design. In the study, 22 volunteer students were assigned to the experimental and control groups by simple randomization. The experimental group was given case-based education to improve their clinical reasoning skills, and the control group continued the standard education process. Data were collected using a Student Information Form, the Clinical Reasoning Case Form (CRCF), the Student Satisfaction with Education Questionnaire, and a Form for Views on the Education. In the evaluation of data, frequency values, Fisher exact test, Mann-Whitney U, and Wilcoxon tests, Cohen's d coefficient for effect size, ITT analysis, and covariance analysis were used.

DETAILED DESCRIPTION:
Aim of the study This study was conducted to determine the effect of case-based education on the development of nursing students' clinical reasoning skills in critical illnesses.

Research hypotheses H01: There is no difference between the experimental group and the control group in terms of their CRCF scores.

H02: Case-based education on clinical reasoning has no positive effect on student satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Having completed the "Medical Nursing" and Surgical Nursing" courses,
* Volunteering to participate in the study,
* Participate in "Case-Based Education"

Exclusion Criteria:

* Not being willing to participate in the study,
* Abandoning the "Case-Based Education" practice
* Not taking one or two of the "Medical Nursing" and "Surgical Nursing" courses at all, or to have taken them but unsuccessfully

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Student Information Form | The measurement was collected one week before education.
  This form consists of 9 questions, including students' nicknames, age, gender, duration of clinical experience, level of school success, and views on the nursing process
Clinical Reasoning Case Form (CRCF) | The first measurement was collected one week before education. The second measurement was collected 3 weeks after education.
  There were 10 clinical cases on the CRCF prepared for the objectives of these three steps in students' clinical reasoning process. The cases involved critical illness, and early warning findings that show worsening in critical illness and are used to determine priority nursing diagnosis.
  Five people, who were experts in the field of medical nursing and had clinical experience, were consulted between February 15 and 28, 2021 to confirm the clinical accuracy and reality of CR cases and their content and comprehensibility. The content validity index of expert opinions evaluated with the Davis technique was determined as 1.

SECONDARY OUTCOMES:
Student Satisfaction with Education Questionnaire | The measurement was collected 3 weeks after education.
  A questionnaire adapted from the study of Lee et al. (2010) was used to evaluate students' satisfaction with the education given. A 6-point Likert-type scale (1= strongly disagree, 6= strongly agree) was used to evaluate the ten items of the questionnaire. The 10th item on the questionnaire is reverse coded. High scores on the questionnaire indicate a high level of satisfaction.
Form for Views on the Education | The measurement was collected 3 weeks after education.
  The effectiveness of the education model was evaluated by the researchers with a SWOT analysis (strengths, weaknesses, opportunities, and threats) based on data collected from students in the experimental group without obtaining nicknames or personal information after the completion of the education via an online questionnaire that consisted of 4 questions about the strengths, weaknesses, perceived threats, and opportunities of the education model.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Nursing, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: Altman, M. R., Kantrowitz-Gordon, I., Moise, E., Malcolm, K., Vidakovic, M., Barrington, W., ... & de Castro, A. B. (2021). Addressing Positionality Within Case-Based Learning to Mitigate Systemic Racism in Health Care. Nurse Educator, 46(5), 284-289. — https://pubmed.ncbi.nlm.nih.gov/33156141/
- See also: Banning, M. (2008). Clinical reasoning and its application to nursing: Concepts and research studies. Nurse education in practice, 8(3), 177-183. — https://pubmed.ncbi.nlm.nih.gov/17869587/
- See also: Dekhtyar, M., Park, Y. S., Kalinyak, J., Chudgar, S. M., Fedoriw, K. B., Johnson, K. J., ... & Stern, S. (2022). Use of a structured approach and virtual simulation practice to improve diagnostic reasoning. Diagnosis, 9(1), 69-76. — https://pubmed.ncbi.nlm.nih.gov/34246202/
- See also: de Sá Tinôco, J. D., Cossi, M. S., & de Carvalho Lira, A. L. B. (2021). Effect of educational intervention on clinical reasoning skills in nursing: A quasi-experimental study. Nurse Educat — https://pubmed.ncbi.nlm.nih.gov/34218071/
- See also: Groves, M., Scott, I., & Alexander, H. (2002). Assessing clinical reasoning: a method to monitor its development in a PBL curriculum. Medical teacher, 24(5), 507-515. — https://pubmed.ncbi.nlm.nih.gov/12450471/
- See also: Hoffman, K. A., Aitken, L. M., & Duffield, C. (2009). A comparison of novice and expert nurses' cue collection during clinical decision-making: Verbal protocol analysis. International journal of nursing studies, 46(10), 1335-1344. — https://pubmed.ncbi.nlm.nih.gov/19555954/
- See also: Hong, S., Lee, J., Jang, Y., & Lee, Y. (2021). A Cross-Sectional Study: What Contributes to Nursing Students' Clinical Reasoning Competence?. International Journal of Environmental Research and Public Health, 18(13), 6833. — https://pubmed.ncbi.nlm.nih.gov/34202159/
- See also: Jacques, T., Harrison, G. A., McLaws, M. L., & Kilborn, G. (2006). Signs of critical conditions and emergency responses (SOCCER): a model for predicting adverse events in the inpatient setting. Resuscitation, 69(2), 175-183. — https://pubmed.ncbi.nlm.nih.gov/16497427/
- See also: Lee, K. C., & Wessol, J. L. (2022). Clinical Reasoning, Judgment, and Safe Medication Administration Practices in Senior Nursing Students. Nurse Educator, 47(1), 51-55. — https://pubmed.ncbi.nlm.nih.gov/34359065/
- See also: Leijser, J., & Spek, B. (2021). Level of clinical reasoning in intermediate nursing students explained by education year and days of internships per healthcare branches: A cross-sectional study. Nurse Education Today, 96, 104641. — https://pubmed.ncbi.nlm.nih.gov/33157365/
- See also: Levett-Jones, T.,... & Hickey, N. (2010). The 'five rights' of clinical reasoning: An educational model to enhance nursing students' ability to identify and manage clinically 'at risk'p — https://pubmed.ncbi.nlm.nih.gov/19948370/
- See also: Ma, C., & Zhou, W. (2022). Effects of unfolding case-based learning on academic achievement, critical thinking, and self-confidence in undergraduate nursing students learning health assessment skills. Nurse Education in Practice, 103321. — https://pubmed.ncbi.nlm.nih.gov/35287002/
- See also: Rohde, E., & Domm, E. (2018). Nurses' clinical reasoning practices that support safe medication administration: An integrative review of the literature. Journal of clinical nursing, 27(3-4), e402-e411. — https://pubmed.ncbi.nlm.nih.gov/28926146/
- See also: Tedesco-Schneck, M. (2019). Use of script concordance activity with the think-aloud approach to foster clinical reasoning in nursing students. Nurse educator, 44(5), 275-277. — https://pubmed.ncbi.nlm.nih.gov/30394999/
- See also: Wong, S. H. V., & Kowitlawakul, Y. (2020). Exploring perceptions and barriers in developing critical thinking and clinical reasoning of nursing students: A qualitative study. Nurse Education Today, 95, 104600. — https://pubmed.ncbi.nlm.nih.gov/32992269/